CLINICAL TRIAL: NCT02903602
Title: Health in the Hands of Women: Test of a Community Health Worker Teaching Method "Sharing Histories"
Brief Title: Sharing Histories: Test of a Teaching Method for Community Health Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future Generations Graduate School (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Instituto de Investigacion Nutricional, Peru (Other)
Responsible Party: Principal Investigator, Laura C. Altobelli, Professor - Principal Investigator, Future Generations Graduate School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FGGS-01; N° AID-OAA-A-10-00048 (Other Grant/Funding Number: US Agency for International Development (USAID))
Record Dates: First submitted 2016-08-31; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infant Nutrition Disorders; Health Behavior
Keywords: sharing histories; autobiographical memory; health behavior; narrative communication; community health workers; global health; maternal and child health; stunting
MeSH Terms: conditions — Infant Nutrition Disorders; Health Behavior; Growth Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHW training method-Sharing Histories (Experimental): Experimental clusters of primary health care facilities provided training to Community Health Workers (CHW) from their communities utilizing the experimental teaching methodology, "Sharing Histories".
  CHW in both study groups made home visits to pregnant women and mothers of children under two years of age to teach mothers, monitor behaviors and danger signs in pregnant women, newborns, and children, and refer cases when needed for preventive and curative care.
  Interventions: Behavioral: Sharing Histories training method for CHW
- CHW training method-Standard (Active Comparator): Control clusters of primary health care facilities provided training to Community Health Workers (CHW) from their communities utilizing a standard CHW teaching methodology.
  CHW in both study groups made home visits to pregnant women and mothers of children under two years of age to teach mothers, monitor behaviors and danger signs in pregnant women, newborns, and children, and refer cases when needed for preventive and curative care.
  Interventions: Behavioral: Standard training method for CHW

INTERVENTIONS:
Behavioral: Sharing Histories training method for CHW — Female Community Health Worker training participants were led through a guided process of recalling and sharing their autobiographical memories of their personal experiences in the first 1000 days of each of their children (pregnancy, childbirth, postpartum, newborn, breastfeeding, complementary feeding, infant diarrhea and hygiene, pneumonia). On the basis of memories, cultural beliefs and practices are identified and training content is built.
  Arms: CHW training method-Sharing Histories
Behavioral: Standard training method for CHW — Female Community Health Workers were trained with standard participatory teaching method with three phases: identify knowledge, provide new knowledge, evaluate learning.
  Arms: CHW training method-Standard

SUMMARY:
The purpose of this study is to determine the effectiveness of an innovative methodology for training Community Health Workers that will improve their effectiveness in educating mothers to adopt best practice health behaviors in the home.

DETAILED DESCRIPTION:
Objective: Training of community health workers (CHW) is a growing priority to close the gap between health services and mothers/families in resource poor communities. To address research needs on how to improve effectiveness of CHW training, the investigators tested an innovative CHW teaching methodology called "Sharing Histories" hypothesizing that this would empower and enable CHW to better teach mothers to improve health knowledge and behaviors that contribute to improved child growth.

Method: The study was a cluster-randomized controlled trial: 22 health facility jurisdictions were matched and randomly assigned as experimental or control. Health personnel Tutors and female CHW were trained using either the "Sharing Histories" methodology (experimental) or a standard but still participatory teaching method (control). Training content, materials, and other interventions were held constant between study groups. Impact on maternal knowledge and practices, and child growth and morbidity were measured in representative household surveys at baseline, midterm, and final evaluation, with 600 mothers interviewed - 300 in each study group - at each point in time.

ELIGIBILITY:
Inclusion Criteria:

* Adult interviewed must be mother or guardian of a child under two years of age.
* Child from birth (0.1 months-old) to under two years of age (23.9 months-old).

Exclusion Criteria:

* If a mother selected for interview had more than one child under age two years, only the younger child was considered for the interview and anthropometry measurements.

Max Age: 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in rate of stunting in children under two years of age (birth to 23.9 months of age) | Chidren born up to 24 months prior to the baseline survey in 2010. Children born up to 24 months prior to the final survey in 2014
  Stunting is defined as low height-for-age less than -2 z-scores from the median on the World Health Organization growth standard, 2006.

CONTACTS AND LOCATIONS:
Overall Officials: Laura C. Altobelli, DrPH, Principal Investigator — Future Generations Graduate School

IPD SHARING:
Plan to Share IPD: Yes
Data set available to researchers by contacting Principal Investigator